CLINICAL TRIAL: NCT05235763
Title: Heart Failure Activity Coach Study
Acronym: HEALTHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CareLigo AB (Industry)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: activity coach
Record Dates: First submitted 2022-01-21; First posted 2022-02-11 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Physical Inactivity; Heart Failure
MeSH Terms: conditions — Sedentary Behavior; Heart Failure

STUDY DESIGN:
Intervention Model Description: Upon recruitment, patients are randomized 1:1 to either intervention or control group. The study arms run in parallell for the twelve weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): A sham activity coach will be installed on the Optilogg system, slightly changing its appearance.
  Interventions: Other: sham activity coach
- Intervention (Experimental): The activity coach educates the patient about physical activity, offers means of manually tracking physical activity, and provides trends of registered activity. Furthermore, it provides weekly summaries of registered physical activity and provides means of setting goals for the following week.
  Interventions: Other: activity coach

INTERVENTIONS:
Other: activity coach — The activity coach educates the patient about physical activity, offers means of manually tracking physical activity, and provides trends of registered activity. Furthermore, it provides weekly summaries of registered physical activity and provides means of setting goals for the following week.
  Arms: Intervention
Other: sham activity coach — The visual appearance of Optilogg is changed as to make the patient aware that something has happened to it, hence not knowing if it is the real activity coach or not. No new functionality is added, however.
  Arms: Control

SUMMARY:
An application (app) called the activity coach will be tested to see if it can increase physical activity and decrease sedentary behaviuor, as well as increase quality of life and lead to personal goal attainment in physically inactive heart failure (HF) patients. This pilot randomized controlled trial (RCT) will test the study design and recruitment process, as well as outcomes for a future efficacy RCT.

HF-patients equipped with the mHealth-tool Optilogg will be screened for physical inactivity and then recruited and randomized to either have the activity coach app added to their Optilogg or remain with the standard Optilogg. The study will go on for 12 weeks. Weeks 1 and 12 physical activity using an accelerometer will be recorded, as well as health-related quality of life. At the start of the study the patients will list goals relating to physical activity which the wish to attain, and the level of attainment will be evaluated at the end of the study.

The activity coach educated the patient about physical activity, offers means of manually tracking physical activity, and provides trends of registered activity. Furthermore, it provides weekly summaries of registered physical activity and provides means of setting goals for the following week.

DETAILED DESCRIPTION:
Study design:

---------------- The activity coach is to be developed using a scientific approach based on the Medical Research Council guidelines, including a small pilot (ethical approval Dnr 2020-01444) which is to be published separately.

This is the first step and the second step is the randomized controlled pilot study (pilot-RCT), to be performed in a primary care setting in Sweden (ethical approval Dnr 2021-05366-01). The purpose is to test the newly developed application (app) called the activity coach, to see if it can improve physical activity, health and quality of life in physically inactive hert failure (HF) patients, but more importantly test the study design and recruitment process, as well as outcomes for a future efficacy RCT.

The patients included will already be equipped with the mHealth tool Optilogg, and then screened for physical inactivty through a self-report question (Blomqvist, 2020, ESC Heart Fail, Utility of single-item questions to assess physical inactivity in patients with chronic heart failure), and then randomized to either receive or not receive the activity coach app.

After randomization the patients will be equipped with an accelerometer for one week. The intervention will go on for 12 weeks, and week twelve the patients will once again carry an acceleroemter.

At baseline demographical data will be recorded, as well as data on co-morbidities and pharmacological treatment. Patients will from a pre-specified list select two goals relating to physical activity that they wish to attain. After 12 weeks they will evaluate the subjective goal attainment on a five level ordinal scale ranging from -2 to 2. At weeks 1 and 12 they will also report health related quality of life using the Kansas City Cardiomyopathy Questionnaire.

Intervention

--------------- The Optilogg system is based around a touch screen computer (tablet), and the activity coach app runs on this screen.

During the first week the patient receives specific education about physical activity and HF on the screen After the first week the patient is expected to be motivated to engage in physical activity and a short slideshow on the screen of the activity coach illustrates how the person using the system can manually register physical activity on the tablet interface. The registered activity trends can be viewed on the screen.At the end of every week the user will receive a weekly summary on screen with the option to set a goal for next week. The goal functionality is optional so that anyone who feels negative stress from the goal, can simply select to not have a goal.

All patients will have access to telephone support during office hours for technical assistance with Optilogg and/or the activity coach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed heart failure
* Equipped with Optilogg
* Physically inactive (screening)

Exclusion Criteria:

* Does not consent to using accelerometer
* Does not consent to home-visit
* Current participation in another study relating to physical activity
* Life-expectancy less than six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Study design | 12 weeks
  Analyze the number of patients needed to be screened to find appropriate and willing participants for the study.

SECONDARY OUTCOMES:
Physical activity | 12 weeks
  Measured with acelerometer, reported as steps per day
Sedentary time | 12 weeks
  Measured with accelerometer, evaluate if sedentary time has been decreased by 10 minutes or more.
Goal attainment score | 12 weeks
  At the start of the study, patients will select to goals relating to physical acitvity which they want to achieve. At the end of the study, this attainment will be evaluated on an ordinal scale with five levels, ranging from -2 to 2, and a mean of the two goal attainments is calculated.
Kansas City Cardiomyopathy Questionnaire | 12 weeks
  Health-related quality of life assessed by Kansas City Cardiomyopathy Questionnaire, a scale between 0 (very poor) to 100 (excellent).

OTHER OUTCOMES:
System adherence | 12 weeks
  For the intervention group, analysis of the frequency with which they used the activity coach

CONTACTS AND LOCATIONS:
Overall Officials: Tiny Jaarsma, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Skiftinge VC, Eskilstuna, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blomqvist A, Back M, Klompstra L, Stromberg A, Jaarsma T. Utility of single-item questions to assess physical inactivity in patients with chronic heart failure. ESC Heart Fail. 2020 Aug;7(4):1467-1476. doi: 10.1002/ehf2.12709. Epub 2020 May 6. PMID 32372549
- [Derived] Blomqvist A, Back M, Klompstra L, Stromberg A, Jaarsma T. Testing the Recruitment Frequency, Implementation Fidelity, and Feasibility of Outcomes of the Heart Failure Activity Coach Study (HEALTHY): Pilot Randomized Controlled Trial. JMIR Form Res. 2025 Jan 8;9:e62910. doi: 10.2196/62910. PMID 39778202
- [Derived] Blomqvist A, Back M, Klompstra L, Stromberg A, Jaarsma T. Usability and feasibility analysis of an mHealth-tool for supporting physical activity in people with heart failure. BMC Med Inform Decis Mak. 2024 Feb 12;24(1):44. doi: 10.1186/s12911-024-02452-z. PMID 38347499